CLINICAL TRIAL: NCT06198998
Title: The Prospective, Multi-center, Single-arm Clinical Evaluation Trial of the CorVad Percutaneous Ventricular Assist System
Brief Title: CorVad Percutaneous Ventricular Assist System Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COREMED_Corvad_HRPCI
Record Dates: First submitted 2023-07-09; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CorVad Percutaneous Ventricular Assist System (Experimental): Subjects with coronary artery disease receiving high-risk PCI will be supported by the CorVad Percutaneous Ventricular Assist System during the procedure.
  Interventions: Device: CorVad Percutaneous Ventricular Assist System

INTERVENTIONS:
Device: CorVad Percutaneous Ventricular Assist System — The CorVad Percutaneous Ventricular Assist System provides hemodynamics support for intraoperative protection during high-risk percutaneous coronary intervention.

SUMMARY:
This study aims to evaluate the safety and effectiveness of the CorVad Percutaneous Ventricular Assist System for short-term ventricular support during high-risk percutaneous coronary intervention (HRPCI) in non-emergent, hemodynamically stable coronary artery disease patients via a prospective, multicenter, single-arm clinical trial.

DETAILED DESCRIPTION:
This prospective, multicentre, single-arm clinical trial of the CorVad Percutaneous Ventricular Assist System is designed to measure the incidence of major adverse cardiovascular and cerebrovascular events (MACCE) at 30 days after PCI and is planned to enrol 120 subjects.

The target population of subjects are patients with coronary artery disease who need high-risk PCI treatment, and sign an informed consent form (ICF) approved by the Ethics Committee (EC). Subjects who meet the enrolment criteria as judged by the investigator will apply the trial product according to the requirements and will be followed up to 30 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years old≤ patient age ≤90 years old;
* 2. Patient willing and able to comply with protocol requirements and data collection procedures; able to understand study purpose and sign informed consent;
* 3. As assessed by the cardiac team the patient needs coronary revascularization, but CABG (Coronary Artery Bypass Grafting) is of high risk, or the patient refuses to undergo CABG. After comprehensive evaluation, the cardiac team believes that the patient can benefit from PCI (Percutaneous Coronary Intervention);
* 4. The patient is hemodynamically stable and meeting one of the following:

  1. Left ventricular ejection fraction (LVEF) ≤30%, with multivessel disease, planning PCI to at least one complex lesion* in a major epicardial vessel or branch;
  2. LVEF ≤35% and either:

     I. Unprotected left main intervention;

     II. Or last patent coronary conduit;
  3. LVEF ≤40%, planning PCI to at least one complex lesion* in a major epicardial vessel or branch. The intervention team confirms there is a risk of cardiac arrest or circulatory collapse. This must be confirmed by at least two associate senior physicians or one chief senior physician.

     * Complex lesions include moderate-to-severe calcification, chronic total occlusions (CTO), diffuse disease, bifurcation lesions, severe tortuosity, etc.

Exclusion Criteria:

* 1. ST-segment elevation myocardial infarction (STEMI) on ECG within 7 days;
* 2. Cardiac arrest requiring cardiopulmonary resuscitation within 24 hours pre-procedure;
* 3. Cardiogenic shock defined as meeting all of the following:

  1. Systolic blood pressure <90mmHg, or requiring vasopressors/inotropes to maintain blood pressure >90mmHg;
  2. Clinical evidence of end-organ hypoperfusion (cold extremities or urine output <30ml/h), or use of IABP or other mechanical circulatory assist device;
  3. Cardiac index (CI) <2.2L/min/m^2 and pulmonary capillary wedge pressure (PCWP) >15mmHg;
* 4. Presence of left ventricular thrombus;
* 5. Presence of mechanical aortic valve or cardiac contractility device;
* 6. Presence of moderate-to-severe aortic valve stenosis;
* 7. Presence of moderate-to-severe aortic valve insufficiency;
* 8. Deemed unable to tolerate percutaneous ventricular assist device based on clinical or imaging assessment, including iliac/femoral artery diameter <6mm, severe tortuosity, severe bilateral iliofemoral/femoral artery disease, or other peripheral vascular disease;
* 9. Presence of aortic vascular disease or aortic dissection;
* 10. Presence of uncorrected, sustained ventricular arrhythmia causing inability to stable position percutaneous ventricular assist device;
* 11. History of stroke with permanent neurological deficit, intracerebral hemorrhage, subdural hematoma, or conditions predisposing to intracranial hemorrhage such as arteriovenous malformation or mass;
* 12. End-stage renal disease requiring dialysis or serum creatinine ≥4mg/dL;
* 13. Presence of potential bleeding diathesis or hypercoagulable state;
* 14. Pregnancy (for women of childbearing potential, pregnancy test required within 7 days prior to PCI procedure);
* 15. Presence of contraindication to anticoagulation;
* 16. History of liver failure, with ALT, AST, and bilirubin elevated to 3 times the upper limit of normal (ULN) or international normalized ratio (INR) ≥2;
* 17. Presence of uncorrected abnormal coagulation parameters (platelet count ≤75,000/mm^3, INR≥2.0, or fibrinogen ≤1.50g/L);
* 18. Presence of uncontrolled active infection requiring antibiotic therapy;
* 19. Participation in any other clinical trial that may impact the results of this study;
* 20. Other circumstances that are unforeseen and determined by the investigator to be unsuitable for the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-10-18 (Estimated); Study Completion 2024-10-18 (Estimated)

PRIMARY OUTCOMES:
Combined incidence of major adverse cardiovascular and cerebrovascular events (MACCE) at 30 days post-PCI. | 30 days post-PCI
  Major adverse events were defined as follows: death, new myocardial infarction, stroke, and target vessel revascularisation.
  Calculation formula:
  30-day MACCE rate = Number of subjects experiencing any MACCE event within 30 days post-PCI ÷ Total number of subjects × 100%

SECONDARY OUTCOMES:
Hemodynamic stability during PCI procedure | During PCI procedure
  Defined as mean arterial pressure (MAP) <60mmHg for no more than 10 minutes during the PCI procedure, without needing additional pharmacological therapy.
PCI procedural angiographic success rate | Post-PCI
  Angiographic success defined as: residual stenosis <30% post stent implantation or residual stenosis <50% post balloon angioplasty. Success rate calculated based on number of treated lesions.
Change of aortic valve regurgitation | Pre-procedure and pre-discharge
  Defined as changing from no or mild aortic regurgitation pre-procedure to moderate or severe regurgitation on pre-discharge echocardiography.
Change in creatinine clearance at 48 hours post-PCI | Pre-procedure and 48 hours post-PCI
  Assessed at 48 hours post-PCI and compared to baseline.
Change in left ventricular ejection fraction (LVEF) pre- and post-PCI | Pre-procedure, 48 hours post-PCI and pre-discharge
  Assessed at 48 hours post-PCI and pre-discharge, and compared to baseline.
Change in New York Heart Association (NYHA) functional classification | Pre-procedure and post-PCI
  Evaluated based on NYHA classification and compared to baseline.
Combined incidence of major adverse cardiovascular and cerebrovascular events (MACCE) at 90 days post-PCI. | 90 days post-PCI
  Major adverse events were defined as follows: death, new myocardial infarction, stroke, and target vessel revascularisation.
  Calculation formula:
  90-day MACCE rate = Number of subjects experiencing any MACCE event within 90 days post-PCI ÷ Total number of subjects × 100%

CONTACTS AND LOCATIONS:
Overall Officials: Ke Fei Dou, Principal Investigator — Cardiometabolic Center, Fuwai Hospital, Chinese Academy of Medical Sciences
Locations (12):
- China (12):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Tangdu Hospital of Air Force Medical University, Xi'an, Shaanxi
  - Shanghai East Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Xijing Hospital of Air Force Military Medical University, Xi’an, Shanxi
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
At this moment the IPD is not yet available for access and will be updated when it is ready.